CLINICAL TRIAL: NCT01938209
Title: A Randomized Control Trial of the Immediate Effects of Seated Thoracic Manipulation and Targeted Supine Thoracic Manipulation on Cervical Spine Flexion Range of Motion and Pain
Brief Title: A Comparison of Seated Thoracic Manipulation and Targeted Supine Thoracic Manipulation on Cervical Flexion Motion and Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chatham University (Other)
Collaborators: Megan J. Olson Hunt (Unknown)
Responsible Party: Principal Investigator, Steve Karas, Assistant Professor, Chatham University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: karas 003; karas thoracic spine
Record Dates: First submitted 2013-09-03; First posted 2013-09-10 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2013-09

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- seated general thoracic spine manipulation (Experimental): seated general thoracic spine manipulation
  Interventions: Other: seated thoracic manipulation
- supine specific thoracic spine manipulation (Experimental): Specific supine manipulation
  Interventions: Other: supine specific thoracic spine manipulation

INTERVENTIONS:
Other: seated thoracic manipulation — seated general thoracic spine manipulation
  Arms: seated general thoracic spine manipulation
Other: supine specific thoracic spine manipulation — supine specific thoracic spine manipulation
  Arms: supine specific thoracic spine manipulation

SUMMARY:
Thirty-nine patients with cervical spine pain were randomly assigned to either a seated thoracic manipulation or targeted supine thoracic manipulation group. Pain and flexion range of motion measures were taken before and after the intervention.

DETAILED DESCRIPTION:
DESIGN: Randomized clinical trial OBJECTIVES: To determine the effectiveness of seated thoracic manipulation versus targeted supine thoracic manipulation on cervical spine pain and flexion range of motion. There is evidence that thoracic spine manipulation is an effective treatment for patients with cervical spine pain. This evidence includes a variety of techniques to manipulate the thoracic spine. While each of them is effective, no research has compared techniques to determine which produces the best outcomes.

METHODS: Thirty-nine patients with cervical spine pain were randomly assigned to either a seated thoracic manipulation or targeted supine thoracic manipulation group. Pain and flexion range of motion measures were taken before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria required patients to be between 18-60 years old with a primary complaint of neck pain

Exclusion Criteria:

* identification of red flags suggestive of nonmusculoskeletal etiology, history of whiplash injury within six weeks of the initial visit, diagnosis of cervical spine stenosis, central nervous system involvement, or signs of nerve root compression (two of the following limited at the same level: strength, sensation, reflexes).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2011-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
neck pain | pain measure taken immediately on first visit
  As measured by patient response at end range of flexion on a scale of 0 - 10.

SECONDARY OUTCOMES:
neck range of motion | range of motion assessed immediately in first visit
  As measure using a bubble goniometer, shich has been shown to be valid and reliable.